CLINICAL TRIAL: NCT03403699
Title: Human iPSC for Repair of Vasodegenerative Vessels in Diabetic Retinopathy
Acronym: iPSC
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Maria Grant, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: 300000173
Record Dates: First submitted 2018-01-11; First posted 2018-01-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Complications; Diabetic Retinopathy
Keywords: inducible pluripotent stem cells
MeSH Terms: conditions — Diabetes Complications; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Inducible pluripotent stem cells will be generated and cryopreserved.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- nondiabetics: Any man or woman between the ages of 21- 98 years of age will be eligible to participate. To participate in the study as a study subject we will require: a) the subject must be a healthy control and b) the subject be willing and have the ability to cooperate with the eye exam and blood draw.
  Interventions: Biological: Generation of inducible pluripotent stem cells
- Diabetic: Any man or woman between the ages of 21- 98 years of age will be eligible to participate. To participate in the study as a study subject we will require: a) carry the diagnosis of diabetes and b) the subject be willing and have the ability to cooperate with the eye exam and blood draw.
  Interventions: Biological: Generation of inducible pluripotent stem cells

INTERVENTIONS:
Biological: Generation of inducible pluripotent stem cells — Generation of inducible pluripotent stem cells from peripheral blood cells.

SUMMARY:
This study proposes to carefully examine the hypothesis that human inducible pluripotent stem cells (iPSCs) can be effectively employed as a future therapeutic option for individuals with diabetic retinopathy and macular ischemia. iPSCs will be generated from the peripheral blood cells of subjects with diabetes and age matched controls. The human iPSC cells will be used to generate mesoderm cells for injection into the vitreous cavity of diabetic rodents and primate eyes. The ability of mesoderm cells to generate endothelial cells and pericytes in areas of degenerated capillaries will be examined. The human iPSCs will also be used to generate hematopoietic CD34+CD45+ cells. The combination of CD34+CD45+ cells derived from iPSCs and iPSC derived mesoderm will be examined in combination for their potentially beneficial effect to enhance the vessel formation.

DETAILED DESCRIPTION:
Vascular complications due to diabetes mellitus (DM) are the result of sustained vascular injury with insufficient vascular repair. In chronic diabetes, vascular reparative mechanism can be lost resulting in development of microvascular complications (MVC), such as diabetic retinopathy (DR). We assessed the reparative function of progenitor cells that circulate in the peripheral blood of diabetic individuals and found that the vascular wall-derived progenitor cells, endothelial colony forming cells (ECFCs), were depleted in diabetics with MVC. Bone marrow-derived progenitor cells, CD45+CD34+ were dysfunctional in diabetics with MVC. We found that human inducible pluripotent stem cells (hiPSCs)-derived ECFCs displayed the ability to form functional and durable blood vessels in vivo and conferred therapeutic revascularization by connecting with and remaining integrated with host rodent vessels long term. We characterized a mesoderm subset (SSEA5-KNA+ cells) generated from hiPSCs that gives rise to ECFCs. Finally, we used hiPSCs to generate CD34+CD45+ cells and tested the impact of co-administration of these cells with ECFCs within the vitreous. The addition of CD34+CD45+ cells with ECFCs resulted in the enhanced survival, function and reparative ability of the ECFCs. This beneficial effect was mediated by reducing retinal oxidative stress and inflammation.

These novel and paradigm shifting findings led us to hypothesize: the hiPSC-derived-mesoderm subset (SSEA5-KNA+) can be utilized for long term revascularization of vasodegenerative capillaries and their reparative action can be further enhanced by coinjection of CD34+CD45+ cells that provide anti-oxidant and anti-inflammatory effects.

ELIGIBILITY:
Inclusion Criteria:

* Any man or woman between the ages of 21- 98 years of age will be eligible to participate. To participate in the study as a study subject we will require: a) the subject must either carry the diagnosis of diabetes or be a healthy aged control and b) the patient be willing and have the ability to cooperate with the eye exam and skin punch biopsy protocol.

Exclusion Criteria:

* We will apply the following exclusion criteria: a) evidence of ongoing acute or chronic infection (HIV, Hepatitis B or C, tuberculosis); b) ongoing malignancy; c) cerebral vascular accident or cerebral vascular procedure; d) current pregnancy; e) history of organ transplantation; f) presence of a graft (to avoid any effect of the graft on inflammatory parameters; and g) patients with anemia. Subjects with AMD, glaucoma, uveitis, known hereditary degenerations or other significant ocular complications other than diabetic retinopathy will be excluded.

Ages: 21 Years to 98 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have retinal abnormalities other than diabetic retinopathy will be excluded. Patients who have history of malignant disease or hematologic disorder. We will record medications that the patient is taking at the time of biopsy. Baseline characteristics will also be recorded, including age, lipid parameters, body mass index, blood pressure, smoking history, antioxidant intake and use of nutritional supplements.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-01-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Generating iPSCs from peripheral blood | From blood draw to 4 months
  Blood will be collected from the patient and cells will be isolated and shipped to ALSTEM for generation of iPSCs
Differentiate iPSCs into CD34+ cells and mesoderm | 4 months to 4 years
  Specific cell culture conditions will be used to differentiate the cells into these two distinct populations

CONTACTS AND LOCATIONS:
Overall Officials: Maria B Grant, MD, Principal Investigator — 1954
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No